CLINICAL TRIAL: NCT01850277
Title: Comparison of a Rhythm Control Treatment Strategy Versus a Rate Control Strategy in Patients With Permanent or Long-term Persistent Atrial Fibrillation and Heart Failure Treated With Cardiac Resynchronization Therapy - a Pilot Study
Brief Title: Cardiac Resynchronization in Atrial Fibrillation Trial - a Pilot Study
Acronym: Pilot-CRAfT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IK-NP-0021-47/1378/13
Record Dates: First submitted 2013-04-22; First posted 2013-05-09 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial fibrillation; Cardiac resynchronization therapy; Heart failure; Rhythm control strategy
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Amiodarone; Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhythm control (Experimental): In this group a strategy to restore and maintain SR, including amiodarone and an external electrical cardioversion (EEC), is implemented. A procedure of AF ablation is possible but not obligatory.
  At baseline, patients assigned to the group undergo a standard 12-lead ECG, a 6-minute walk test (6MWT), a cardiopulmonary exercise test(CPX), an echocardiography(ECHO), a standard device control; a serum thyroid -stimulating hormone (TSH) level is assessed and patients fill the Minnesota Living With Heart Failure Questionnaire (MLHFQ). Control visits are performed every 3 months including a 12-lead ECG measurement and a device control. On the visits in the 3rd and 12th month an ECHO, a CPX, a 6MWT are performed and a MLHFQ is filled; control TSH levels are assessed every 6 months.
  Interventions: Drug: Amiodarone; Procedure: External electrical cardioversion (EEC)
- Rate control (Active Comparator): In the latter group a pharmacotherapy to slow and control ventricular rate by means of pharmacotherapy and an atrio-ventricular junction ablation (AVJA) is implemented.
  At baseline, each patient assigned to the rate control group undergoes a standard 12-lead ECG, a 6MWT, a CPX, an ECHO, a standard device control and a serum TSH level assessed. Moreover, the patient fills the Minnesota Living With Heart Failure Questionaire (MLHFQ). The control visits are performed for one year, every 3 months including a standard 12-lead ECG measurement and standard control of the device. On the visits in the 3rd and 12th month additionally an ECHO, a CPX, a 6MWT are performed and a MLHFQ is filled. The control TSH levels are assessed every 6 months.
  Interventions: Drug: Pharmacotherapy to slow and control ventricular rate; Procedure: Atrioventricular junction ablation (AVJA)

INTERVENTIONS:
Drug: Amiodarone — The pharmacological treatment in the rhythm control strategy consist of amiodarone given orally including the loading dose up to 600mg daily - for the first 4 weeks. Then, a maintenance dose of 200mg/daily is prescribed. The use of other anti-arrhythmic agents is possible unless they are contraindicated. The introduction of amiodarone must not be performed unless the patient is treated effectively with oral anticoagulants for 3 weeks at least. Discontinuation of amiodarone results neither in withdrawal from the study nor in change of the treatment arm.
  Other Names: Cordarone; Amiodaron; Pacerone; Aratac; Cardinorm; Rithmik; Arycor; Atlansil; Tachyra
  Arms: Rhythm control
Procedure: External electrical cardioversion (EEC) — The first EEC is performed after the loading dose of amiodarone has been administered. A maximal number of shocks during one cardioversion is 3. The amount of the energy delivered during shocks is left at discretion of a physician performing the EEC. The EEC must be performed in accordance with the present guidelines on EEC and post-procedural care and the state of art.
  If atrial fibrillation reoccur, the patient should undergo a next EEC as soon as possible but preserving the safety time margins (i.e. effective anticoagulation period). The maximal no. of EEC procedures is 3. If sinus rhythm resumption or its maintenance is impossible or AF reoccur after the 3rd EEC, a strategy of rhythm control is discontinued and a rate control strategy is implemented.
  Arms: Rhythm control
Drug: Pharmacotherapy to slow and control ventricular rate — The pharmacotherapy should be consistent with current guidelines. It should include negative chronotropic and negative dromotropic agents such as beta-blockers, digitalis and amiodarone (the use of other, less popular agents, is also possible). The choice of the agents as well as their dosages are left at discretion of the treating physician. The goal of the therapy is to obtain BiVp% >95%
  Other Names: beta-blockers; digitalis; amiodarone
  Arms: Rate control
Procedure: Atrioventricular junction ablation (AVJA) — The procedure of atrioventricular junction ablation is dedicated to the patients in the rate control group in who the rate control is unsatisfactory. An AVJA procedure is not obligatory. The decision to perform an AVJA should be discussed with the patient and should be made collectively by the therapeutic team.
  Arms: Rate control

SUMMARY:
The purpose of this prospective randomized study is to determine whether patients on cardiac resynchronization therapy with concomitant long-standing persistent or permanent atrial fibrillation would benefit from a strategy to restore and maintain sinus rhythm (rhythm control strategy) in comparison to a rate control strategy in terms of higher biventricular paced beats percentage.

DETAILED DESCRIPTION:
Due to a lack of sufficient data the present guidelines on treatment of patients with atrial fibrillation (AF) and cardiac resynchronization therapy (CRT) devices are of low scientific evidence. The efficacy of CRT in AF patients is limited by the percentage of the effective biventricular paced beats (BiVp%), which should exceed 95%-98% - a goal which is seldom obtained by means of pharmacological rate control strategy. The only treatment strategy which effect is scientifically established is an atrioventricular junction ablation (AVJA) but the use of this method is limited.

On the other hand, about 10% of patients with persistent forms of AF experience a spontaneous sinus rhythm (SR) resumption after CRT implantation. Moreover, SR resumption and it's maintenance by means of single external electrical cardioversion in AF patients has been proven feasible. A strategy of rhythm control in AF patients on CRT could provide high BiVp% and improve the efficacy of CRT in this group of patients.

To show superiority of the rhythm control strategy over the rate control strategy a sample size of 60 patients was calculated based on following assumptions: two-tailed test, a type I error of 0.05, a power of 80%, efficacy (mean BiVp%) of rate control strategy 90%, efficacy (mean BiVp%)of rhythm control strategy 98% and 8% drop-out rate to fulfill the criteria of intention-to-treat analysis. Due to presumed lack of statistical power the secondary end points and safety endpoints will be considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Permanent or long-standing persistent atrial fibrillation (definitions according to the latest European Society of Cardiology guidelines on AF)
* At least 3 months after a procedure of a CRT device implantation
* A CRT device with a presence of a right atrial electrode
* Age: ≥18 years old
* Effectively biventricular paced captured beats <95%
* Effective therapy with oral anticoagulants for at least 3 months
* Written informed consent

Exclusion Criteria:

* Reversible causes of AF
* Significant valve disease
* Advanced A-V block (including: AVJA)
* Contraindications to amiodarone (hyperthyroidism, not compensated hypothyroidism, drug intolerance, QT>460ms for men, QT>450 for women)
* Long-QT syndrome
* Decompensation of the heart failure within 48 hours before the qualification
* Cardiac transplantation in 6 months
* Life expectancy less than 1 year
* Chronic dialysis
* LA diameter >6cm
* Alcohol abuse
* Pregnancy/lack of effective contraceptive therapy (in case of females in the reproductive age)
* Participation in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
BiVp% | 1 year
  Percentage of effective biventricular paced beats during 1st year (mean percentage from baseline to the control visit in 12th month) .

SECONDARY OUTCOMES:
6MWT distance | 1 year
  6 minute walk test distance (in meters)measured at 1 year from baseline
peak VO2 | 1 year
  Peak oxygen uptake (peak VO2) measured by means of cardiopulmonary exercise test at 1 year from baseline
NYHA class | 1 year
  Heart failure (HF) symptoms escalation measured in New York Heart Association (NYHA) classes at 1 year from baseline
Ejection fraction | 1 year
  Ejection fraction (EF) [%] assessed in ECHO at 1 year from baseline
LVEDD reduction from baseline at 1 year | baseline and 1 year
  Change from baseline in left ventricle end-diastolic diameter (LVEDD) in ECHO at 1 year
LVEDV reduction from baseline at 1 year | baseline and 1 year
  Change from baseline in left ventricle end-diastolic volume (LVEDV) in ECHO at 1 year
LVESD reduction from baseline at 1 year | baseline and 1 year
  Change from baseline in left ventricle end-systolic diameter (LVESD) in ECHO at 1 year
LVESV reduction froma baseline at 1 year | baseline and 1 year
  Change from baseline in left ventricle end-systolic volume (LVESV) in ECHO at 1 year
Reduction of LA diameter at 1 year | baseline and 1 year
  Change from baseline in left atrium diameter assessed in ECHO at 1 year
Reduction of mitral regurgitation at 1 year | baseline and 1 year
  Change from baseline in mitral regurgitation measured in ECHO at 1 year
Heart failure exacerbations | up to 1 year
  Number of heart failure exacerbations in the treatment arm in 1 year time from baseline
Mortality | up to 1 year
  Numer of deaths assesed in 1 year follow-up
Stroke/TIA | up to 1 year
  Stroke or transient ischemic attack (TIA) during a year follow-up
CV mortality | up to 1 year
  Death due to cardiovascular (CV) causes during a year follow-up
Cardiovascular hospitalizations | up to 1 year
  Number of hospitalizations due to cardiovascular causes during a year follow-up
Quality of Life | 1 year
  The quality of life measured with the Minnesota Living with Heart Failure Questionaire (MLHFQ) at 1 year from baseline
AF prevalence | 1 year
  Measurement of the prevalence of atrial fibrillation (precentage of participants with AF) at 1 year from baseline
Ventricular arrhythmia | up to 1 year
  Number of ventricular arrhythmias (VF/"Torsade de Pointes" VT/sVT/nsVT) during the first year from basline
Electrotherapy | up to 1 year
  The number of high-energy interventions ("shocks") including separately: adequate shocks, inadequate shocks, electrical storm applies only to the patients with CRT-D device during the first year from baseline
Side effects | 1 year
  Overall number of side effects cases and complications cases of the treatment strategies related to: the device, the pharmacotherapy, the electrotherapy during the first year from baseline.
6MWT distance | 3 months
  6 minute walk test distance (in meters) at 3 months from baseline
peak VO2 | 3 months
  Peak oxygen uptake (peak VO2) measured by means of cardiopulmonary exercise test at 3 months from baseline
NYHA class | 3 months
  Heart failure (HF) symptoms escalation measured in New York Heart Association (NYHA) classes at 3 months from baseline
Ejection fraction | 3 months
  Ejection fraction (EF) [%] assessed in ECHO at 3 months from baseline
LVEDD reduction | baseline and 3 months
  Change from baseline in left ventricle end-diastolic diameter (LVEDD) reduction in ECHO at 3 months
LVEDV reduction | baseline and 3 months
  Change from baseline in left ventricle end-diastolic volume (LVEDV) reduction in ECHO at 3 months
Reduction of LA area | baseline and 1 year
  Change from baseline in left atrium area assessed in ECHO at 1 year
Reduction of LA diameter | baseline and 3 months
  Change from baseline in left atrium diameter assessed in ECHO at 3 months
Reduction of mitral regurgitation | baseline and 3 months
  Change from baseline in mitral regurgitation measured in ECHO at 3 months
Stroke/TIA | up to 3 months
  Stroke or transient ischemic attack (TIA) during the first 3 months from baseline
Quality of Life | 3 months
  The quality of life measured with the Minnesota Living with Heart Failure Questionaire (MLHFQ) at 3 months from baseline
BiVp% | 3 months
  Percentage of effective biventricular paced beats during first 3 months from baseline.
AF prevalence | 3 months
  Measurement of the prevalence of atrial fibrillation (precentage of participants with AF) at 3 month from baseline
Electrotherapy | up to 3 months
  The number of high-energy interventions ("shocks") including separately: adequate shocks, inadequate shocks, electrical storm applies only to the patients with CRT-D device during first 3 months from baseline
Ventricular arrhythmia | up to 3 months
  Number of ventricular arrhythmias (VF/"Torsade de Pointes" VT/sVT/nsVT) during the first 3 months from basline
Side effects | 3 months
  Overall number of cases of side effects and complications of the treatment strategies related to: device, pharmacotherapy, electrotherapy during the first 3 months from baseline.
Reduction of LA area | baseline and 3 month
  Change from baseline in left atrium area assessed in ECHO at 3 months

OTHER OUTCOMES:
Identification of the factors predicting the response to the rhythm control strategy | 1 year
  Identification of the patients which benefit the most from the rhythm control strategy and comparison of their baseline characteristics with the whole group. Identification of non-responders to the rhythm control strategy and comparison of their baseline characteristics with the whole group. (multiple regression analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Jan B Ciszewski, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Maciej Sterlinski, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, II Dept. of Coronary Heart Disease, Warsaw, Poland

REFERENCES:
- [Derived] Ciszewski JB, Tajstra M, Kowalik I, Maciag A, Chwyczko T, Jankowska A, Smolis-Bak E, Firek B, Zajac D, Karwowski J, Szwed H, Pytkowski M, Gasior M, Sterlinski M. Rhythm and rate control strategies in patients with long-standing persistent atrial fibrillation treated with cardiac resynchronization: the results of the randomized Pilot-CRAfT study. Clin Res Cardiol. 2024 Oct 10. doi: 10.1007/s00392-024-02541-z. Online ahead of print. PMID 39387937
- [Derived] Ciszewski J, Maciag A, Kowalik I, Syska P, Lewandowski M, Farkowski MM, Borowiec A, Chwyczko T, Pytkowski M, Szwed H, Sterlinski M. Comparison of the rhythm control treatment strategy versus the rate control strategy in patients with permanent or long-standing persistent atrial fibrillation and heart failure treated with cardiac resynchronization therapy - a pilot study of Cardiac Resynchronization in Atrial Fibrillation Trial (Pilot-CRAfT): study protocol for a randomized controlled trial. Trials. 2014 Oct 4;15:386. doi: 10.1186/1745-6215-15-386. PMID 25281275